CLINICAL TRIAL: NCT00170339
Title: Bone Density and Serum Testosterone in Male Methadone Maintained Patients
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Other Study IDs: HSR-04-2404; 0409M63575
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Opiate Dependence; Osteoporosis; Erectile Dysfunction; Hypogonadism
Keywords: Opiate Dependence; Methadone Maintenance; Osteoporosis; Hypogonadism
MeSH Terms: conditions — Opioid-Related Disorders; Osteoporosis; Erectile Dysfunction; Hypogonadism

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a pilot study designed to answer the question " Do men who are receiving methadone maintenance therapy have lower spinal bone densities compared with age-matched controls who are not receiving methadone therapy?"

The primary aim is to assess whether the mean or median spinal dual-ray energy x-ray absorptiometry (DEXA) scan results are different between these two groups of male patients. Primary measurements include: spinal bone densitometry by DEXA scan.

The secondary aim is to examine the role of sex steroids in men receiving methadone maintenance therapy and their association with spinal bone density and sexual dysfunction. Secondary measurements include: serum testosterone, estradiol, lutenizing hormone, albumin, sex hormone binding globulin and Vitamin D levels; age; Brief Sexual Function Inventory; Dietary, smoking/alcohol use and physical activity; Medical history, surgical and medication use; length of time using illicit opiates and time on methadone maintenance therapy.

DETAILED DESCRIPTION:
Chronic use of opiates has long been associated with multiple side effects, many of which are due to lower levels of androgens in this patient population. Previous studies have shown that long-term opiate use may lead to narcotic induced hypogonadism, resulting in significantly decreased testosterone levels in men. One area of chronic opiate use that has not been looked at extensively is the correlation between narcotic-induced hypogonadism and associated side effects such as osteoporosis and sexual dysfunction in male patients receiving methadone maintenance therapy. Marked testosterone deficiency is a well-established rick factor for both osteoporosis and altered sexual function, and recent information demonstrated that altered estrogen levels may play a role in these side effects as well. Thre present pilot study investigates the role of sex steroids in male patients maintained on methadone therapy and their association with bone densitometry and sexual dysfunction. Free testosterone, estradiol, lutenizing hormone, sex hormone binding globulin, Vitamin D levels and albumin will be measured in thirty community-dwelling outpatient men participating in a methadone maintenance program as well as thirty age-matched controls from a general medicine clinic. Osteodensitometry will be performed with the DEXA technique at the lumbar spine. Participants will also complete the Brief Male Sexual Function Inventory as well as be assessed for smoking/alcohol use, calcium intake, physical activity, length of time receiving opiates as well as concurrent medications. It is hypothesized that patients receiving methadone maintenance therapy will have lower bone mass densities, free testosterone, estradiol, and sexual dysfunction scores than the age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 50
* methadone maintenance for at least 12 months (for cases)
* stable dose of methadone for 6 months (for cases)
* willing to participate in the study
* competency in English
* male

Exclusion Criteria:

* previous diagnosis of sexual dysfunction
* previous diagnosis of osteoporosis
* serum creatinine > 2 mg/dL
* chronic opiate use (for controls)
* congestive heart failure
* illicit drug use

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2005-04; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Wesa, M.D., Principal Investigator — Hennepin Faculty Associates/ Hennepin County Medical Center
Locations (1):
- Hennepin Faculty Associates/ Hennepin County Medical Center, Minneapolis, Minnesota, United States